CLINICAL TRIAL: NCT02380573
Title: Cognitive and Functional Connectivity Effects of Methylene Blue in Healthy Aging, Mild Cognitive Impairment and Alzheimer's Disease
Brief Title: Effects of Methylene Blue in Healthy Aging, Mild Cognitive Impairment and Alzheimer's Disease
Acronym: MB2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Texas Alzheimer's Research and Care Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC20150410H
Record Dates: First submitted 2015-02-24; First posted 2015-03-05 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Mild Cognitive Impairment; MCI; Aging; Alzheimer's Disease; AD
Keywords: methylene blue; fMRI
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Methylene Blue; Indigo Carmine; Phenazopyridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Healthy Aging MB (Experimental): Methylene Blue (USP grade, 282mg oral, daily, 2 weeks, 12 weeks) Phenazopyridine hydrochloride (97.5 mg oral, 2 weeks, 12 weeks)
  Interventions: Drug: Methylene Blue; Drug: Phenazopyridine hydrochloride
- Healthy Aging Placebo (Placebo Comparator): Drug: FD&C Blue # 2 (USP grade, 282 mg oral, 2 weeks, 12 weeks) Phenazopyridine hydrochloride (97.5 mg oral, 2 weeks, 12 weeks)
  Interventions: Drug: FD&C Blue # 2; Drug: Phenazopyridine hydrochloride
- Mild Cognitive Impairment (MCI) MB (Experimental): Methylene Blue (USP grade, 282 mg oral, daily, 2 weeks, 12 weeks) Phenazopyridine hydrochloride (97.5 mg oral, 2 weeks, 12 weeks)
  Interventions: Drug: Methylene Blue; Drug: Phenazopyridine hydrochloride
- Mild Cognitive Impairment (MCI) Placebo (Placebo Comparator): Drug: FD&C Blue # 2 (USP grade, 282 mg oral, 2 weeks, 12 weeks) Phenazopyridine hydrochloride (97.5 mg oral, 2 weeks, 12 weeks)
  Interventions: Drug: FD&C Blue # 2; Drug: Phenazopyridine hydrochloride
- Mild Alzheimer's Disease (AD) MB (Experimental): Methylene Blue (USP grade, 282 mg oral, daily, 2 weeks, 12 weeks) Phenazopyridine hydrochloride (97.5 mg oral, 2 weeks, 12 weeks)
  Interventions: Drug: Methylene Blue; Drug: Phenazopyridine hydrochloride
- Mild Alzheimer's Disease (AD) Placebo (Placebo Comparator): Drug: FD&C Blue # 2 (USP grade, 282 mg oral, 2 weeks, 12 weeks) Phenazopyridine hydrochloride (97.5 mg oral, 2 weeks, 12 weeks)
  Interventions: Drug: FD&C Blue # 2; Drug: Phenazopyridine hydrochloride
- Healthy Middle Age MB (Experimental): Methylene Blue (USP grade, 282 mg oral, daily, 2 weeks, 12 weeks) Phenazopyridine hydrochloride (97.5 mg oral, 2 weeks, 12 weeks)
  Interventions: Drug: Methylene Blue; Drug: Phenazopyridine hydrochloride
- Healthy Middle Age Placebo (Placebo Comparator): Drug: FD&C Blue # 2 (USP grade, 282 mg oral, 2 weeks, 12 weeks) Phenazopyridine hydrochloride (97.5 mg oral, 2 weeks, 12 weeks)
  Interventions: Drug: FD&C Blue # 2; Drug: Phenazopyridine hydrochloride

INTERVENTIONS:
Drug: Methylene Blue
  Other Names: Phenothiazin-5-ium, 3, 7-bis (dimethylamino)-chloride, trihydrate
  Arms: Healthy Aging MB; Healthy Middle Age MB; Mild Alzheimer's Disease (AD) MB; Mild Cognitive Impairment (MCI) MB
Drug: FD&C Blue # 2
  Other Names: Placebo
  Arms: Healthy Aging Placebo; Healthy Middle Age Placebo; Mild Alzheimer's Disease (AD) Placebo; Mild Cognitive Impairment (MCI) Placebo
Drug: Phenazopyridine hydrochloride
  Other Names: Azo

SUMMARY:
A double-blind, placebo-controlled study that aims to investigate the effect of 2-week and 12-week administration of USP methylene blue (MB) on cerebral blood flow, functional connectivity, memory and attention cognitive abilities using fMRI and behavioral measures in healthy aging, mild cognitive impairment (MCI) and mild Alzheimer's disease (AD) subjects.

DETAILED DESCRIPTION:
Healthy aging and aging human subjects with mild cognitive impairment and mild Alzheimer's disease from the TARCC cohort and South Texas will be studied using a double-blind, placebo-controlled design. After informed consent and familiarity with the tasks and the MRI environment, the subject will enter an MRI scanner and perform the following 6 tasks.

fMRI and behavioral data will be collected simultaneously while inside the scanner.

Delayed match-to-sample task: The subject views a pattern for a few seconds and then is prompted to recall the memorized pattern using a response system (approx. 10 mins).

Face-name task: The subject is shown blocks of stimuli where a novel or familiar face is paired with a name. In a later run, the subjects are asked whether the correct name is matched with the correct face. (approx. 10 mins).

Psychomotor vigilance task: The subject receives a visual cue that alerts them to press a button as fast as possible. (approx. 10 mins).

Cerebral Blood Flow and Resting State fMRI: Subject scanned with eyes closed and told to not think about a particular topic, each lasting about 10 minutes.

fMRI data acquisition: fMRI and neuropsychological battery measurements will be made before the intervention. These measurements will then be repeated after 2 weeks and 12 weeks.

fMRI will image changes in regional brain activity associated with these tasks. The MRI pulse sequences include diffusion tensor imaging, standard and non-invasive anatomical and quantitative MRI for coregistration and blood-oxygen-level dependent (BOLD) fMRI.

CO2 challenge: Cerebral blood flow measurements will be obtained while the subject rests in the scanner after administration of medical-grade 5% CO2 in air for 3-5 minutes. This will be repeated on weeks 2 and 12.

Data analysis: Standard fMRI analysis will be analyzed using established fMRI software. Statistical parametric analysis will be performed to generate activation maps. fMRI data will be corrected for multiple comparisons using a false discovery rate (q < 0.05) and threshold for cluster values to conservatively control for type I error. Behavioral data will be analyzed with paired t-test and ANOVA calculations used for group comparison with p < 0.05 (with Bonferroni correction) considered statistically significant.

Expected results: The investigators predict that, compared to placebo, MB will: i) improve working memory retention in a delayed match-to-sample task by memory performance and enhanced fMRI responses in the prefrontal cortex and parietal lobes, ii) improve episodic memory as determined by fMRI activation in the hippocampus, medial temporal lobes and prefrontal cortex iii) reduce reaction time in a psychomotor vigilance test and enhance fMRI responses within a cortical sustained attention network iv) improve CBF and v) improve fMRI connectivity in default mode and visuospatial and memory networks/subnetworks. The fMRI and behavioral performance effects on memory will be greater in the MCI and mild AD groups than in the healthy aging group. The effects will be greater in the MCI and AD groups than in the control groups.

Power analysis: Sample sizes were calculated using an fMRI power tool based on pilot data from the current study for a power of 80%, alpha = 0.05, False Discovery Rate < 0.05, to detect statistical difference between MB and placebo23. The investigators estimate they will need 20-25 subjects per arm of group (complete studies) and thus will recruit 200-240 subjects to account for potential failed studies.

ELIGIBILITY:
Inclusion Criteria for all subjects:

1. 45-89 years old
2. All genders
3. All minorities
4. English, Spanish, or multilingual speakers
5. Postmenopausal or surgically sterile females only.
6. Inclusion for MCI group only: participants will meet the criteria for amnestic and non-amnestic MCI such as those currently used by Texas Alzheimer's Research and Care Consortium (TARCC) consensus diagnosis
7. Inclusion for AD group only: Alzheimer's Early-stage, sporadic-type

Exclusion Criteria:

1. Pregnancy or breastfeeding
2. Contraindication for MRI (Claustrophobia and magnetic metal implants)
3. Glucose-6-phosphate deficiency, methemoglobinemia
4. Allergy to MB
5. Color-blindness
6. Craniotomy, craniectomy or endovascular neurosurgery
7. A current diagnosis of stroke, transient ischemic attack (TIA), any primary neurodegenerative disorder, or any other causes of neuropsychologic disturbances or secondary dementia (MCI or AD does not exclude subject)
8. A serious intercurrent illness likely to cause death within the next 5 years, such as terminal cancer
9. Alcohol and/or drug abuse
10. Any detection of an unknown disease process (eg. new tumor) on the study's neuroimaging at the discretion of the investigators
11. A systolic blood pressure ≥180 mmHg and/or a diastolic blood pressure ≥105 mmHg
12. Severe difficulty or an inability to perform any one of the 6 Katz Activities of Daily Living
13. Patients who are unlikely to comply with trial visit schedule or with trial medication,
14. On any psychiatric serotonergic antidepressant medication or psychotropic medication within the last 5 weeks
15. Diagnosis of epilepsy, traumatic brain injury with loss of consciousness, psychosis, panic attacks,
16. Chronic kidney disease, cirrhosis, liver or renal transplants
17. Known hypersensitivity to thiazide diuretics and phenothiazines
18. Any other condition, which in the opinion of the investigator, would put the participant at risk and warrant exclusion from the study

Ages: 45 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2015-07; Primary Completion 2022-04-21 (Actual); Study Completion 2023-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Imaging Institute, The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

REFERENCES:
- [Background] Bruchey AK, Gonzalez-Lima F. Behavioral, Physiological and Biochemical Hormetic Responses to the Autoxidizable Dye Methylene Blue. Am J Pharmacol Toxicol. 2008 Jan 1;3(1):72-79. doi: 10.3844/ajptsp.2008.72.79. PMID 20463863
- [Background] Rojas JC, Bruchey AK, Gonzalez-Lima F. Neurometabolic mechanisms for memory enhancement and neuroprotection of methylene blue. Prog Neurobiol. 2012 Jan;96(1):32-45. doi: 10.1016/j.pneurobio.2011.10.007. Epub 2011 Nov 3. PMID 22067440
- [Background] Telch MJ, Bruchey AK, Rosenfield D, Cobb AR, Smits J, Pahl S, Gonzalez-Lima F. Effects of post-session administration of methylene blue on fear extinction and contextual memory in adults with claustrophobia. Am J Psychiatry. 2014 Oct;171(10):1091-8. doi: 10.1176/appi.ajp.2014.13101407. PMID 25018057
- [Background] Lin AL, Poteet E, Du F, Gourav RC, Liu R, Wen Y, Bresnen A, Huang S, Fox PT, Yang SH, Duong TQ. Methylene blue as a cerebral metabolic and hemodynamic enhancer. PLoS One. 2012;7(10):e46585. doi: 10.1371/journal.pone.0046585. Epub 2012 Oct 9. PMID 23056355
- [Background] Huang S, Du F, Shih YY, Shen Q, Gonzalez-Lima F, Duong TQ. Methylene blue potentiates stimulus-evoked fMRI responses and cerebral oxygen consumption during normoxia and hypoxia. Neuroimage. 2013 May 15;72:237-42. doi: 10.1016/j.neuroimage.2013.01.027. Epub 2013 Jan 26. PMID 23357077
- [Background] Talley Watts L, Long JA, Chemello J, Van Koughnet S, Fernandez A, Huang S, Shen Q, Duong TQ. Methylene blue is neuroprotective against mild traumatic brain injury. J Neurotrauma. 2014 Jun 1;31(11):1063-71. doi: 10.1089/neu.2013.3193. Epub 2014 Apr 8. PMID 24479842
- [Background] Long JA, Watts LT, Chemello J, Huang S, Shen Q, Duong TQ. Multiparametric and longitudinal MRI characterization of mild traumatic brain injury in rats. J Neurotrauma. 2015 Apr 15;32(8):598-607. doi: 10.1089/neu.2014.3563. Epub 2015 Jan 22. PMID 25203249
- [Background] Rodriguez P, Jiang Z, Huang S, Shen Q, Duong TQ. Methylene blue treatment delays progression of perfusion-diffusion mismatch to infarct in permanent ischemic stroke. Brain Res. 2014 Nov 7;1588:144-9. doi: 10.1016/j.brainres.2014.09.007. Epub 2014 Sep 8. PMID 25218555
- [Background] Shen Q, Du F, Huang S, Rodriguez P, Watts LT, Duong TQ. Neuroprotective efficacy of methylene blue in ischemic stroke: an MRI study. PLoS One. 2013 Nov 21;8(11):e79833. doi: 10.1371/journal.pone.0079833. eCollection 2013. PMID 24278191
- [Background] Peter C, Hongwan D, Kupfer A, Lauterburg BH. Pharmacokinetics and organ distribution of intravenous and oral methylene blue. Eur J Clin Pharmacol. 2000 Jun;56(3):247-50. doi: 10.1007/s002280000124. PMID 10952480
- [Background] Gonzalez-Lima F, Bruchey AK. Extinction memory improvement by the metabolic enhancer methylene blue. Learn Mem. 2004 Sep-Oct;11(5):633-40. doi: 10.1101/lm.82404. PMID 15466319
- [Background] Naylor GJ, Martin B, Hopwood SE, Watson Y. A two-year double-blind crossover trial of the prophylactic effect of methylene blue in manic-depressive psychosis. Biol Psychiatry. 1986 Aug;21(10):915-20. doi: 10.1016/0006-3223(86)90265-9. PMID 3091097
- [Background] Mackworth JF. Vigilance, arousal, and habituation. Psychol Rev. 1968 Jul;75(4):308-22. doi: 10.1037/h0025896. No abstract available. PMID 4875885
- [Background] Rombouts SA, Barkhof F, Goekoop R, Stam CJ, Scheltens P. Altered resting state networks in mild cognitive impairment and mild Alzheimer's disease: an fMRI study. Hum Brain Mapp. 2005 Dec;26(4):231-9. doi: 10.1002/hbm.20160. PMID 15954139
- [Background] Wang L, Li H, Liang Y, Zhang J, Li X, Shu N, Wang YY, Zhang Z. Amnestic mild cognitive impairment: topological reorganization of the default-mode network. Radiology. 2013 Aug;268(2):501-14. doi: 10.1148/radiol.13121573. Epub 2013 Mar 12. PMID 23481166
- See also: Texas Alzheimer's Research and Care Consortium — http://www.txalzresearch.org
- See also: Research Imaging Institute — http://ric.uthscsa.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Aging MB: Methylene Blue (USP grade, 282mg oral, daily, 2 weeks, 12 weeks) Phenazopyridine hydrochloride (97.5 mg oral, 2 weeks, 12 weeks)
  Methylene Blue
  Phenazopyridine hydrochloride
- Healthy Aging Placebo; Mild Cognitive Impairment (MCI) Placebo; Mild Alzheimer's Disease (AD) Placebo; Healthy Middle Age Placebo: Drug: FD&C Blue # 2 (USP grade, 282 mg oral, 2 weeks, 12 weeks) Phenazopyridine hydrochloride (97.5 mg oral, 2 weeks, 12 weeks)
  FD&C Blue # 2
  Phenazopyridine hydrochloride
- Mild Cognitive Impairment (MCI) MB; Mild Alzheimer's Disease (AD) MB; Healthy Middle Age MB: Methylene Blue (USP grade, 282 mg oral, daily, 2 weeks, 12 weeks) Phenazopyridine hydrochloride (97.5 mg oral, 2 weeks, 12 weeks)
  Methylene Blue
  Phenazopyridine hydrochloride
Period: Overall Study
Arm/Group | Healthy Aging MB | Healthy Aging Placebo | Mild Cognitive Impairment (MCI) MB | Mild Cognitive Impairment (MCI) Placebo | Mild Alzheimer's Disease (AD) MB | Mild Alzheimer's Disease (AD) Placebo | Healthy Middle Age MB | Healthy Middle Age Placebo
Started | 22 | 21 | 28 | 24 | 1 | 2 | 0 | 0
Completed | 12 | 13 | 12 | 16 | 1 | 1 | 0 | 0
Not Completed | 10 | 8 | 16 | 8 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Because this was a study of aging people, participants under the age of 18 were not included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Aging MB | Healthy Aging Placebo | Mild Cognitive Impairment (MCI) MB | Mild Cognitive Impairment (MCI) Placebo | Mild Alzheimer's Disease (AD) MB | Mild Alzheimer's Disease (AD) Placebo | Healthy Middle Age MB | Healthy Middle Age Placebo | Total
Number analyzed (Participants) | 22 | 21 | 28 | 24 | 1 | 2 | 0 | 0 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 6 | 4 | 0 | 0 | 0 | 0 | 17
  >=65 years | 19 | 17 | 22 | 20 | 1 | 2 | 0 | 0 | 81
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 17 | 18 | 1 | 1 | 0 | 0 | 58
  Male | 9 | 13 | 11 | 6 | 0 | 1 | 0 | 0 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White, Non-Hispanic | 11 | 11 | 7 | 6 | 1 | 2 |  |  | 38
  Race/Ethnicity: White, Hispanic | 11 | 8 | 18 | 16 | 0 | 0 |  |  | 53
  Race/Ethnicity: Pacific Islander, Non-Hispanic | 0 | 0 | 0 | 0 | 0 | 0 |  |  | 0
  Race/Ethnicity: Pacific Islander, Hispanic | 0 | 0 | 1 | 0 | 0 | 0 |  |  | 1
  Race/Ethnicity: Black, Non-Hispanic | 0 | 1 | 1 | 0 | 0 | 0 |  |  | 2
  Race/Ethnicity: Black, Hispanic | 0 | 0 | 0 | 1 | 0 | 0 |  |  | 1
  Race/Ethnicity: Asian, Non-Hispanic | 0 | 0 | 0 | 1 | 0 | 0 |  |  | 1
  Race/Ethnicity: Asian, Hispanic | 0 | 0 | 0 | 0 | 0 | 0 |  |  | 0
  Race/Ethnicity: White, Not Specified | 0 | 1 | 0 | 0 | 0 | 0 |  |  | 1
  Race/Ethnicity: Not Specified, Not Specified | 0 | 0 | 1 | 0 | 0 | 0 |  |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 22 | 21 | 28 | 24 | 1 | 2 |  |  | 98

OUTCOME MEASURES:

1. Primary Outcome: fMRI Measurement
Description: fMRI measurement of task blocked activation during Wechsler Memory Scale III
Time Frame: baseline, 2 weeks and 12 weeks
Population: There was not sufficient data collected to be analyzed for Mild Alzheimer's disease MB or placebo, only the scale score was measured, as reported in the Wechsler Memory Scale outcome.
Measure: Mean (Standard Deviation); unit: voxels
Groups:
- Mild Alzheimer's Disease MB: Methylene Blue (USP grade, 282 mg oral, daily, 2 weeks, 12 weeks) Phenazopyridine hydrochloride (97.5 mg oral, 2 weeks, 12 weeks)
- Mild Alzheimer's Disease Placebo: Drug: FD&C Blue # 2 (USP grade, 282 mg oral, 2 weeks, 12 weeks) Phenazopyridine hydrochloride (97.5 mg oral, 2 weeks, 12 weeks)
Arm/Group | Healthy Aging MB | Healthy Aging Placebo | Mild Cognitive Impairment (MCI) MB | Mild Cognitive Impairment (MCI) Placebo | Mild Alzheimer's Disease MB | Mild Alzheimer's Disease Placebo
Number analyzed (Participants) | 12 | 13 | 12 | 16 | 0 | 0
voxels
  Baseline | 2267.0 (2428.23) | 1491.23 (1343.81) | 673.31 (1366.69) | 989.19 (1651.97) |  |
  2 weeks | 1719.00 (1377.02) | 962.69 (843.93) | 12270.59 (1955.60) | 930.25 (1157.55) |  |
  12 weeks | 1451.83 (1623.84) | 1623.84 (919.08) | 1238.58 (1743.67) | 1334.38 (2341.44) |  |

2. Primary Outcome: Wechsler Memory Scale, Third Edition
Description: Working memory task behavioral measures (ie. correct number of responses) Score is 0-104, with higher scores being better.
Time Frame: baseline, 2 weeks ± 3 days, 12 weeks ± 3 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Aging MB | Healthy Aging Placebo | Mild Cognitive Impairment (MCI) MB | Mild Cognitive Impairment (MCI) Placebo | Mild Alzheimer's Disease (AD) MB | Mild Alzheimer's Disease (AD) Placebo
Number analyzed (Participants) | 12 | 14 | 13 | 15 | 1 | 1
score on a scale
  baseline | 14.58 (2.35) | 15.43 (2.85) | 15.23 (2.5) | 13.06 (3.23) | 4 (0) | 15 (0)
  2 weeks | 16 (2.3) | 17.29 (1.33) | 15.23 (2.68) | 15.31 (2.94) | 5 (0) | 17 (0)
  12 weeks | 15.58 (2.11) | 15.93 (2.13) | 14.69 (1.55) | 13.2 (3.17) | 11 (0) | 13 (0)

3. Primary Outcome: fMRI During FNAME
Description: Functional Magnetic Resonance Imaging (fMRI) measurement of task blocked activation.
  Measure reflects blood flow counts, and is not a scale with a high or low score.
Time Frame: baseline, 2 weeks ± 3 days,12 weeks ± 3 days
Population: There was not sufficient data collected to be analyzed for Mild Alzheimer's disease MB or placebo, only the scale measure was obtained in the next outcome.
Measure: Mean (Standard Deviation); unit: voxels activated over a threshold
Groups:
- Healthy Middle Age Placebo: FD&C Blue # 2 (USP grade, 282 mg oral, 2 weeks, 12 weeks) Phenazopyridine hydrochloride (97.5 mg oral, 2 weeks, 12 weeks)
Arm/Group | Healthy Aging MB | Healthy Aging Placebo | Mild Cognitive Impairment (MCI) MB | Mild Cognitive Impairment (MCI) Placebo | Mild Alzheimer's Disease (AD) MB | Mild Alzheimer's Disease (AD) Placebo | Healthy Middle Age MB | Healthy Middle Age Placebo
Number analyzed (Participants) | 12 | 13 | 12 | 16 | 1 | 1 | 0 | 0
voxels activated over a threshold
  baseline | 16881.03 (8823.60) | 17382.29 (6401.56) | 13166.23 (4796.32) | 13777.75 (8955.52) | 2211.00 (0) | 3938.00 (0) |  |
  2 weeks | 18146.92 (7075.66) | 19748.86 (8221.18) | 12935.15 (7042.78) | 15617.31 (7519.81) | 4939.00 (0) | 4140.00 (0) |  |
  12 weeks | 16893.83 (6689.61) | 18342.57 (8230.30) | 13973.56 (10759.77) | 14466.56 (9944.16) | 2240.00 (0) | 1355.00 (0) |  |

4. Primary Outcome: FNAME
Description: Face-Name Task behavioral measures (ie. correct recalls). The FNAME is a cross-modal associative memory test which includes 16 face-name pairs and 16 face-occupation pairs, with a total of 32 pairs to remember. Scores range from 0-32, higher scores are better
Time Frame: baseline, 2 weeks ± 3 days,12 weeks ± 3 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Aging MB | Healthy Aging Placebo | Mild Cognitive Impairment (MCI) MB | Mild Cognitive Impairment (MCI) Placebo | Mild Alzheimer's Disease (AD) MB | Mild Alzheimer's Disease (AD) Placebo
Number analyzed (Participants) | 12 | 14 | 13 | 16 | 1 | 1
score on a scale
  baseline | 14.5 (4.83) | 14.36 (4.86) | 10.54 (3.71) | 11.19 (4.23) | 8 (0) | 6 (0)
  2 weeks | 16.08 (4.7) | 15.36 (6.1) | 12.54 (4.52) | 11.5 (4.62) | 2 (0) | 9 (0)
  12 weeks | 16.67 (4.16) | 16 (6.24) | 14 (3.96) | 12.69 (5.62) | 6 (0) | 1 (0)

5. Primary Outcome: fMRI During Psychomotor Vigilance Task
Description: fMRI measurement of task blocked activation
Time Frame: baseline,2 weeks ± 3 days,12 weeks ± 3 days
Population: There was no data collected to be analyzed for Mild Alzheimer's disease MB or placebo.
Measure: Mean (Standard Deviation); unit: # voxels beyond a threshold
Groups:
- Mild Alzheimer's Disease Placebo: FD&C Blue # 2 (USP grade, 282 mg oral, 2 weeks, 12 weeks) Phenazopyridine hydrochloride (97.5 mg oral, 2 weeks, 12 weeks)
Arm/Group | Healthy Aging MB | Healthy Aging Placebo | Mild Cognitive Impairment (MCI) MB | Mild Cognitive Impairment (MCI) Placebo | Mild Alzheimer's Disease MB | Mild Alzheimer's Disease Placebo
Number analyzed (Participants) | 12 | 13 | 12 | 16 | 0 | 0
# voxels beyond a threshold
  baseline | 271.33 (590.79) | 150.79 (348.98) | 145.00 (321.47) | 56.94 (220.91) |  |
  2 weeks | 175.08 (370.05) | 129.00 (230.28) | 89.54 (173.65) | 75.31 (148.86) |  |
  12 weeks | 66.25 (94.43) | 47.43 (105.62) | 156.77 (330.64) | 13.88 (38.76) |  |

6. Primary Outcome: Psychomotor Vigilance Task
Description: Psychomotor vigilance task (PVT) behavioral measures (ie. reaction time). The primary outcome measures of PVT performance, lapses, are defined as reaction times exceeding 500 msec or failure to react. The PVT lapses are believed to represent perceptual, processing, or executive failures in the central nervous system (CNS) Lower scores are better, as they indicate quicker reaction times.
Time Frame: baseline, change from baseline at 2 weeks ± 3 days, change from baseline at 12 weeks ± 3 days
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Healthy Aging MB | Healthy Aging Placebo | Mild Cognitive Impairment (MCI) MB | Mild Cognitive Impairment (MCI) Placebo | Mild Alzheimer's Disease (AD) MB | Mild Alzheimer's Disease (AD) Placebo
Number analyzed (Participants) | 12 | 13 | 12 | 16 | 1 | 1
milliseconds
  baseline | 399.9 (58.5) | 382.7 (39.6) | 408.1 (99) | 482.4 (134.5) | 744.8 (0) | 631.04 (0)
  2 weeks | 390.1 (48.85) | 371.86 (47.56) | 402.3 (66.15) | 456.03 (132.94) | 629 (0) | 618.83 (0)
  12 weeks | 397.5 (62.9) | 365.33 (43.53) | 390.7 (80.72) | 455.3 (131.5) | 524.7 (0) | 695.05 (0)

7. Primary Outcome: Wechsler Memory Scale III, Logical Memory Subset
Description: The patient is read two stories, out loud, by the test administrator. After each story is read, the patient is then asked to tell the story back to the administrator, as well as possible. Scores range from 0-75, with higher scores indicating better outcome.
Time Frame: baseline, then 12 weeks ± 3 days
Population: Not all participants came back for all three visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Aging MB | Healthy Aging Placebo | Mild Cognitive Impairment (MCI) MB | Mild Cognitive Impairment (MCI) Placebo | Mild Alzheimer's Disease (AD) MB | Mild Alzheimer's Disease (AD) Placebo
Number analyzed (Participants) | 20 | 19 | 21 | 21 | 1 | 1
score on a scale
  baseline | 47 (9.5) | 43.5 (9.5) | 32.4 (9.66) | 37.48 (9.8) | 25 (0) | 5 (0)
  12 weeks: number analyzed (Participants) | 12 | 13 | 16 | 12 | 1 | 1
  12 weeks | 48 (10.1) | 41.1 (9.1) | 33.5 (7.9) | 37.06 (7.7) | 21 (0) | 5 (0)

8. Primary Outcome: Mini-Mental State Exam (MMSE)
Description: Short screening tool for providing an overall measure of cognitive impairment in clinical, research and community settings. The MMSE contains 11 questions with scores ranging from 1-5 depending on how many responses are required for each question. One point is assigned for each correct answer. The total score can range from 0-30 with a higher score indicating better cognitive skills.
Time Frame: baseline, 2 weeks ± 3 days,12 weeks ± 3 days
Population: Not all participants returned for all three visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Aging MB | Healthy Aging Placebo | Mild Cognitive Impairment (MCI) MB | Mild Cognitive Impairment (MCI) Placebo | Mild Alzheimer's Disease (AD) MB | Mild Alzheimer's Disease (AD) Placebo
Number analyzed (Participants) | 22 | 21 | 28 | 24 | 1 | 2
score on a scale
  baseline: number analyzed (Participants) | 21 | 19 | 21 | 21 | 1 | 2
  baseline | 29 (1.05) | 29.32 (.95) | 27.76 (1.9) | 27.52 (1.86) | 21 (0) | 21 (0)
  3 weeks: number analyzed (Participants) | 21 | 19 | 21 | 21 | 1 | 2
  3 weeks | 29.7 (.66) | 29.6 (.61) | 28.3 (1.15) | 27.7 (2.4) | 26 (0) | 20 (0)
  12 weeks: number analyzed (Participants) | 12 | 13 | 16 | 12 | 1 | 2
  12 weeks | 29.9 (.58) | 29.3 (1.11) | 28.5 (1.4) | 28.25 (1.1) | 24 (0) | 24 (0)

9. Primary Outcome: CLOX: An Executive Clock Drawing Test
Description: The subject draws a clock that says 1:45. Performance is rated according to the CLOX directions, and scored as "CLOX1" with scores ranging from 0-15 with a lower score indicating greater impairment. CLOX1 reflects performance in a novel and ambiguous situation. The CLOX's second step is a simple copying task. The examiner allows the patient to observe him or her drawing a clock in the circle provided on the scoring sheet. The examiner sets the hands again to "1:45", places the 12, 6, 3, and 9 first, and makes the hands into arrows. The patient is allowed to copy the examiner's clock. This clock is scored as "CLOX2" with scores ranging from 0-15 with a lower score indicating greater impairment. Participants can earn up to 15 points for each test, this is summed to give a possible score out of 30 with a higher score indicating less cognitive impairment. Scores reported are from inter-rater reliability
Time Frame: baseline, 2 weeks ± 3 days, 12 weeks ± 3 days
Population: It was determined after the study began that recruiting middle aged subjects would not be worthwhile.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Aging MB | Healthy Aging Placebo | Mild Cognitive Impairment (MCI) MB | Mild Cognitive Impairment (MCI) Placebo | Mild Alzheimer's Disease (AD) MB | Mild Alzheimer's Disease (AD) Placebo
Number analyzed (Participants) | 22 | 21 | 28 | 24 | 1 | 2
score on a scale
  baseline: number analyzed (Participants) | 21 | 19 | 21 | 21 | 1 | 2
  baseline | .89 (.96) | 1 (1.33) | 1.86 (1.85) | 1.52 (1.72) | 1 (0) | 1 (0)
  2 weeks: number analyzed (Participants) | 21 | 19 | 21 | 21 | 1 | 2
  2 weeks | .6 (.75) | .68 (1) | 0.571 (0.978) | -0.857 (1.77) | 2 (0) | 7 (0)
  12 weeks: number analyzed (Participants) | 12 | 13 | 16 | 12 | 1 | 2
  12 weeks | .67 (.63) | .69 (1.6) | 1 (1.13) | .86 (1.54) | 3 (0) | 4 (0)

10. Secondary Outcome: Cerebral Blood Flow Measures
Description: Resting measurements will be used to assess response and CBF using fMRI. Scores are baseline, percent change between baseline and 2 weeks, baseline and 12 weeks
Time Frame: baseline, 2 weeks ± 3 days, 12 weeks ± 3 days
Measure: Mean (Standard Deviation); unit: percentage of change
Groups:
- AD MB: Methylene Blue (USP grade, 282mg oral, daily, 2 weeks, 12 weeks) Phenazopyridine hydrochloride (97.5 mg oral, 2 weeks, 12 weeks)
  Methylene Blue
  Phenazopyridine hydrochloride
- AD Placebo: Drug: FD&C Blue # 2 (USP grade, 282 mg oral, 2 weeks, 12 weeks) Phenazopyridine hydrochloride (97.5 mg oral, 2 weeks, 12 weeks)
  FD&C Blue # 2
  Phenazopyridine hydrochloride
Arm/Group | Healthy Aging MB | Healthy Aging Placebo | Mild Cognitive Impairment (MCI) MB | Mild Cognitive Impairment (MCI) Placebo | AD MB | AD Placebo
Number analyzed (Participants) | 12 | 13 | 12 | 16 | 1 | 1
percentage of change
  baseline | 34.65 (15.62) | 37.9 (49) | 31.97 (16) | 35.2 (35) | 95.13 (0) | 4.02 (0)
  % change, baseline vs 2 weeks | 36.1 (22.9) | 35.97 (27.3) | 31.97 (16) | 31.55 (14.84) | 35.85 (0) | 23.93 (0)
  % change, baseline vs 12 weeks | 40.89 (29) | 42.13 (32.6) | 57.07 (64.1) | 35.2 (14.85) | -1.91 (0) | 48.57 (0)

11. Other Pre Specified Outcome: Functional Connectivity Measures
Description: Functional magnetic resonance imaging (fMRI) measurements will be obtained while the subject rests in the scanner, with their eyes closed. The default mode network (DMN) will be identified from the resting state data using temporal concatenation independent components analysis. Dual regression will then be applied to identify the individual subject's DMN maps, followed by the counting of significant voxels above threshold within the DMN masks. This will be repeated on weeks 2 and 12. the voxel is a 3-dimensional unit that embeds the signals in brain scans. As the MRI machine scans through each dimension of the brain millimeter by millimeter, voxels are formed to enclose the signals created by protons-magnet interactions.
Time Frame: baseline, 2 weeks ± 3 days, 12 weeks ± 3 days
Measure: Mean (Standard Deviation); unit: Voxels
Arm/Group | Healthy Aging MB | Healthy Aging Placebo | Mild Cognitive Impairment (MCI) MB | Mild Cognitive Impairment (MCI) Placebo | Mild Alzheimer's Disease (AD) MB | Mild Alzheimer's Disease (AD) Placebo
Number analyzed (Participants) | 12 | 13 | 12 | 16 | 1 | 1
Voxels
  baseline | 4703.08 (735.81) | 4314.29 (943.58) | 4811.23 (834.89) | 4980 (1809.93) | 3819 (0) | 2990 (0)
  2 weeks | 4778.42 (563.19) | 4066.14 (1392.99) | 5053.38 (956.65) | 4504.81 (1671.78) | 5672 (0) | 3566 (0)
  12 weeks | 4862.75 (730.38) | 4197.64 (1662.41) | 5124.92 (984.09) | 4804.81 (1128.53) | 4541 (0) | 2006 (0)

12. Other Pre Specified Outcome: CO2 Challenge
Description: Cerebral blood flow measurements will be acquired during a brief (3-5 minutes) inhalation of medical-grade 5% CO2 in air. Cerebral blood flow measurements will be obtained using Arterial Spin Labeling (ASL) during a brief (3-5 minutes) inhalation of medical-grade 5% CO2 in air. Mean regional CBF (rCBF) in gray matter is quantified as ml/100g/min of tissue. The percent change from baseline will be calculated. This will be repeated on weeks 2 and 12.
Time Frame: baseline, change from baseline at 2 weeks ± 3 days, change from baseline at 12 weeks ± 3 days
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Healthy Aging MB | Healthy Aging Placebo | Mild Cognitive Impairment (MCI) MB | Mild Cognitive Impairment (MCI) Placebo | Mild Alzheimer's Disease (AD) MB | Mild Alzheimer's Disease (AD) Placebo
Number analyzed (Participants) | 12 | 14 | 13 | 16 | 1 | 1
percentage change from baseline
  baseline | 34.65 (15.62) | 37.90 (49.03) | 31.97 (16.04) | 35.23 (34.99) | 95.13 (0) | 4.02 (0)
  2 weeks | 36.10 (22.95) | 35.97 (27.30) | 29.22 (24.47) | 31.55 (14.85) | 35.85 (0) | 23.93 (0)
  12 weeks | 40.89 (29.05) | 42.13 (32.85) | 57.07 (64.10) | 35.19 (20.83) | -1.91 (0) | 48.57 (0)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of randomization to 12 weeks
Groups:
- Mild Alzheimer's Disease (AD) Placebo: FD&C Blue # 2 (USP grade, 282 mg oral, 2 weeks, 12 weeks) Phenazopyridine hydrochloride (97.5 mg oral, 2 weeks, 12 weeks)
Arm/Group | Healthy Aging MB | Healthy Aging Placebo | Mild Cognitive Impairment (MCI) MB | Mild Cognitive Impairment (MCI) Placebo | Mild Alzheimer's Disease (AD) MB | Mild Alzheimer's Disease (AD) Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21 | 0/28 | 0/24 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21 | 0/28 | 0/24 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 22/22 | 19/21 | 27/28 | 21/24 | 0/1 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Aging MB (N=22) | Healthy Aging Placebo (N=21) | Mild Cognitive Impairment (MCI) MB (N=28) | Mild Cognitive Impairment (MCI) Placebo (N=24) | Mild Alzheimer's Disease (AD) MB (N=1) | Mild Alzheimer's Disease (AD) Placebo (N=1)
blue or orange urine (Renal and urinary disorders) | 22 | 18 | 25 | 20 | NA | NA — blue or orange urine
green stool (Gastrointestinal disorders) | 12 | 14 | 10 | 13 | NA | NA — stool turned green
urinary frequency or urgency (Renal and urinary disorders) | 12 | 2 | 4 | 5 | NA | NA — increased urinary frequency
vomiting or nausea (Gastrointestinal disorders) | 6 | 4 | 7 | 1 | NA | NA — vomiting or nausea
diarrhea/loose stool (Gastrointestinal disorders) | 2 | 6 | 3 | 5 | NA | NA — diarrhea or loose stool
hot flashes (General disorders) | 0 | 0 | 1 | 0 | NA | NA — flashes of heat
bladder irritation (Renal and urinary disorders) | 7 | 0 | 6 | 1 | NA | NA — irritation of bladder
leg cramps (Musculoskeletal and connective tissue disorders) | 4 | 1 | 8 | 1 | NA | NA — leg cramps
decreased libido (Social circumstances) | 1 | 0 | 0 | 0 | NA | NA — decreased in libido
fever (General disorders) | 1 | 0 | 0 | 0 | NA | NA — fever
skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | NA | NA — skin problems

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT02380573/Prot_SAP_000.pdf